CLINICAL TRIAL: NCT07332013
Title: Non-invasive Evaluation of Urinary Titin as an IND-enabling Biomarker for Use in Duchenne Muscular Dystrophy (DMD) Clinical Trials
Brief Title: Urinary Titin Biomarker in DMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-021450; U01NS134672 (NIH)
Record Dates: First submitted 2025-11-06; First posted 2026-01-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Duchenne Muscular Dystrophy (DMD); Becker's Muscular Dystrophy (BMD)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Descending stair walk

INTERVENTIONS:
Other: Descending stair walk — Subjects will participate in a brief on-site, descending stair walk. Subjects will walk down stairs, up to a maximum 2 floors, under the supervision of a physical therapist or study team member.

SUMMARY:
A universal challenge in clinical investigation of novel therapeutics is the need for quantitative, objective biomarkers that directly address the mechanisms of disease and provide information relevant to clinically meaningful functional improvement. This has been a particular challenge in rare and slowly progressive diseases such as Duchenne Muscular Dystrophy (DMD).

The investigators hypothesize that urinary N-terminal fragment of titin (NTFT) corresponding to activity level/intensity will define a high-precision, non-invasive biomarker of systemic muscle injury to enable serial measurements of efficacy and safety in the clinical investigation of gene therapy for DMD and other myopathies. This should provide a valuable exploratory, secondary and eventually primary outcome measure of therapeutic efficacy to minimize the enrollment size in informative early phase and pivotal clinical trials.

DETAILED DESCRIPTION:
The investigators are recruiting ambulatory individuals with Duchenne Muscular Dystrophy (DMD) or Becker Muscular Dystrophy (BMD), and healthy volunteers.

At 3 regular clinical visits, participants will perform a descending stair walk down 2 flights of stairs. Urine will be collected before and after to measure how urinary N-terminal fragment of titin (NTFT) levels are impacted by the activity. Participants will also perform a standard battery of neuromuscular tests, including North Star Ambulatory Assessment and Timed Function Tests. These will be performed as part of the regular clinic visit. Participants will wear an activity monitor during all tests.

After both the first and second visits, participants will be sent home with an activity monitor to measure the participants activity over the course of 7 days. The participant's urine will be collected and frozen 3 times a day (morning, afternoon, and evening) during this period. The investigators will correlate physical activity intensity with the urinary NTFT (titin) levels and the severity of the disease (which will be based on the results of clinical neuromuscular tests).

If there is a clinically-indicated blood draw, participants will have the option to allow collection of an additional sample for exploratory analysis of additional biomarkers.

ELIGIBILITY:
DMD/BMD Subject Inclusion/Exclusion Criteria

Inclusion Criteria:

1. Ambulatory at screening
2. Genetically confirmed diagnosis of DMD/BMD
3. Parental/guardian permission (informed consent) for children. Child assent will also be obtained from patients ages 7 years old and older and deemed by the investigator to be neurodevelopmentally appropriate
4. Access to electricity and a freezer in the home, in order to utilize the provided device and store collected samples

Exclusion Criteria:

* Non-ambulatory at Screening, defined as unable to walk independently and needing assistive devices
* Female patients
* Parental/guardian unable to provide informed consent

Healthy Control Subject Inclusion/Exclusion Criteria

Inclusion criteria:

1. Healthy children without DMD, BMD, or other significant chronic medical disease
2. Ambulatory at Screening, defined as able to walk independently without assistive devices
3. Parental/guardian permission (informed consent). Child assent will also be obtained from patients aged 7 years and older and deemed by the investigator to be neurodevelopmentally appropriate.
4. Access to electricity and a freezer in the home, in order to utilize the provided device and store collected samples

Exclusion criteria:

* Non-ambulatory at Screening, defined as unable to walk independently and needing assistive devices
* Female patients
* Parental/guardian unable to provide informed consent

Ages: 2 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in urinary NTFT (titin) after structured activity | Day 1, 6-12 months , 12-18 months
  Change in urinary NTFT concentration will be measured before and after clinical visits, during which subjects will complete standard of care physical therapy assessments and perform a two-flight stair descent (if able).
Urinary NTFT (titin) relative during unstructured activity in home environment | Day 1, 6-12 months, 12- 18 months
  Change in urinary NTFT (titin) concentration over 1 week in response to unstructured activity at home and will be measured after each scheduled visit. This period of home NTFT monitoring will occur at the same time as activity monitoring described in outcome measure #3.
Unstructured activity level as assessed by wearable activity device | Day 1, 6-12 months, 12-18 months
  Subjects' daily movement and activity levels will be measured continuously over 1 week at home using a pair of wearable accelerometry sensors. This will be completed after each scheduled clinical visit. This period of home activity monitoring will occur in conjunction with NTFT monitoring as described in outcome measure #2.

SECONDARY OUTCOMES:
Change in neuromuscular performance over time, as assessed by routine North Star Ambulatory Assessment (NSAA) | Day 1, 6-12 months, 12-18 months
  North Star Ambulatory Assessment is a standardized set of 17 different activities such as standing, sitting, climbing up and down one step, getting up from the floor, walking, and balancing, which will measure the subjects' motor function while the PT assesses their performance. NSAA will be evaluated at each scheduled visit. The change over time will be evaluated.
Neuromuscular performance over time, as assessed by time to rise from floor (TTR). | Day 1, 6-12 months, and 12-18 months
  The time it takes the participant to get up from the floor will be evaluated at each scheduled visit. The change in TTR over time will be evaluated.
Neuromuscular performance over time, as assessed by 4 stair climb (4SC). | Day 1, 6-12 months, 12-18 months
  The time it takes the participant to climb 4 stairs will be evaluated at each scheduled visit. The change in 4SC over time will be evaluated.
Neuromuscular performance over time, as assessed by 10 meter walk (10MW) | Day 1, 6-12 months, 12-18 months
  The time it takes the participant to walk 10 meters will be evaluated at each scheduled visit. The change in 10MW time over time will be evaluated.
Types of activities | Day 1, 6-12 months, 12-18 months
  Subject's will record type of activity and time spent doing activities in an activity log. The amount of time spent doing activities involving walking and running will be quantified for each study group during 1 week at home following each scheduled visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Yum, MD, Principal Investigator — Children's Hospital of Philadelphia; Benjamin Kozyak, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No